CLINICAL TRIAL: NCT00816257
Title: Lung Transplant Specimen Repository and Data Registry Protocol
Status: Completed | Type: Observational
Sponsor: Karen Wood (Other)
Responsible Party: Sponsor-Investigator, Karen Wood, Karen Wood M.D., Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2005H0101
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Lung Transplantation
Keywords: lung tissue repository

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BAL specimen blood lung biopsy specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
All patients enrolled in the registry will be recipients of single and double lung transplantation (bilateral sequential, heart-lung, or living related donor grafts). During the routine management of lung recipients frequent surveillance of the lung allograft is necessary. This routinely involves: measurement of pulmonary functions, chest radiography, collection of peripheral blood to assess other organ function and monitor therapeutic drug levels, and bronchoscopic evaluation allowing for collection of lung lavage fluid and lung tissue biopsy. This surveillance normally follows a set schedule during the first one to two years following the transplant procedure. Surveillance is routinely performed at weeks 2, 8, 12, 24, 36, and 52 during the first year following the transplant procedure. Additional surveillance may be performed at any time when clinically indicated for the optimal management of the recipient. Information and specimens collected from each of these encounters will be entered in the data registry and specimen repository.

DETAILED DESCRIPTION:
The collection of disposable lung allograft (transplant tissue samples), blood samples and information from medical records for storage, future analysis and research. Stored samples will be available to other researchers who have obtained separate review and approval from an ethics committee called an Institutional Review Board.

Immediately prior to the transplant surgery, the surgeon or pulmonologist will routinely examine the lungs via bronchoscopy during which subjects will be medicated for pain.

The samples that are obtained during this and post-surgery (clinically scheduled) bronchoscopies, including bronchial lavage, are either sent to pathology or are discarded if they do not qualify to go to pathology. For this research, the researchers are asking that the samples that do not qualify for pathology be placed into the repository instead of being thrown away.

ELIGIBILITY:
Inclusion Criteria:

* recipients of single and double lung transplantation (bilateral sequential, heart-lung, or living related donor grafts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2005-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
data registry and lung tissue repository | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: David Nunley, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States